CLINICAL TRIAL: NCT00635479
Title: Role of Vacuum Assisted Closure (VAC) Device in Postoperative Management of Pelvic and Acetabular Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of California, Davis (Other); University of Alabama at Birmingham (Other); Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Brett Crist, Assistant Professor, Co-Director of Trauma Services, Co-Director Trauma Fellowship, Department of Orthopaedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 1096320; 1138438
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Pelvic Fractures; Acetabular Fractures; Hip Fractures
Keywords: Fractures; Pelvic bones; Acetabulum; Hip bones
MeSH Terms: conditions — Hip Fractures; Fractures, Bone | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VAC Device placement (Experimental): will have the VAC device used for post-operative management of acetabular fractures and pelvic fractures.
  Interventions: Device: VAC device
- Gauze dressing (Active Comparator): will receive current traditional surgical wound management with daily dressing changes in post operative management of acetabular fractures and pelvic fractures.
  Interventions: Other: Gauze dressing

INTERVENTIONS:
Device: VAC device — Vacuum Assisted Closure (VAC) device for surgical incision
  Other Names: Wound Vac; Negative pressure wound therapy (NPWT); Incisional Vac
  Arms: VAC Device placement
Other: Gauze dressing — Gauze dressing for surgical incision
  Arms: Gauze dressing

SUMMARY:
The purpose of this research is to study the efficacy and cost effectiveness of the VAC device in comparison to traditional gauze wound dressing in pelvic, acetabular and hip fractures, specifically to see if there is a reduction in the incidence of post operative surgical wound drainage, infections, and hospital stay.

DETAILED DESCRIPTION:
Soft tissue injuries are commonly associated with pelvic and acetabular injuries and additional tissue injury occurs during surgery. Post operative wound drainage, infections and prolonged hospital stay are a common problem during postoperative care. Traditional treatment is dressing of the surgical wound with different conventional dressings.

Use of negative pressure wound therapy has been shown to be beneficial in significantly decreasing wound drainage. Stannard et al. reported the results of randomizing 44 patients with lower extremity fractures (including 4 pilon fractures) into either receiving standard post operative dressing versus NPWT (negative pressure wound therapy). His results showed no difference in infection rate or wound breakdown, but did show a significant difference in the drainage time. The NPWT group stopped draining 3 days earlier than the standard dressing group. The use of NPWT has greatly increased over the years and has been an important adjunct to wound management. These results and anecdotal clinical experience with the use of NPWT (wound VAC) has led us to develop our research question; Does the use of incisional VAC following pelvic &/or acetabular surgery decrease wound complications.

The VAC (KCI USA) device is relatively new device that utilizes negative pressure as a treatment modality for soft tissue injuries following high velocity injuries. VAC device exerts intermittent or constant negative pressure and removes excess fluid from the interstitial space and increases perfusion through vessels. Previous VAC studies showed decreased bacterial load after applying VAC device to the infected wounds.

There have been no randomized studies to prove the cost effectiveness and efficacy of VAC device in reducing wound drainage, infections, and prolonged hospital stays in comparison to traditional gauze dressing wound management during post operative management of pelvic and acetabular fractures.

In examining the incidence of wound complications/infections, we can determine if the incisional VAC decreases the need for additional intervention and if there are any patient related factors (i.e. obesity) related to increased risk of wound complications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Scheduled for surgical repair of pelvic and/or acetabular fracture
* Subject/guardian able to provide informed consent

Exclusion Criteria:

* Less than 18 years of age
* Subject/guardian unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2008-03; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett D Crist, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- VAC Device: Vacuum Assisted Closure (VAC) device
  Wound Vac: Vacuum Assisted Closure (VAC) device for surgical incision
- Gauze Dressing: Gauze Dressing
  Gauze dressing: Gauze dressing for surgical incision
Period: Overall Study
Arm/Group | VAC Device | Gauze Dressing
Started | 55 | 60
Completed | 49 | 42
Not Completed | 6 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAC Device | Gauze Dressing | Total
Number analyzed (Participants) | 55 | 60 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (19.6) | 48.3 (20.1) | 47.6 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 31
  Male | 43 | 41 | 84
Region of Enrollment [Number; unit: participants]
  United States | 55 | 60 | 115

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Infections
Time Frame: Until wound healed, up to 1 year
Measure: Number; unit: participants
Arm/Group | VAC Device | Gauze Dressing
Number analyzed (Participants) | 49 | 42
participants | 5 | 2

ADVERSE EVENTS:
Arm/Group | VAC Device | Gauze Dressing
Serious Adverse Events (participants affected / at risk) | 15/49 | 9/42
Other Adverse Events (participants affected / at risk) | 3/49 | 5/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAC Device (N=49) | Gauze Dressing (N=42)
infection (Infections and infestations) | 10 | 4
Perforated colon (Gastrointestinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
CVA (Vascular disorders) | 0 | 1
implant failure (Surgical and medical procedures) | 2 | 1
prescription overdose (General disorders) | 1 | 0
DVT (Vascular disorders) | 0 | 1
PE (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAC Device (N=49) | Gauze Dressing (N=42)
urinary tract infection (Renal and urinary disorders) | 0 | 2
ileus (Gastrointestinal disorders) | 1 | 0
Regional Pain Syndrome (Nervous system disorders) | 0 | 1
pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
hematoma (Vascular disorders) | 1 | 0
malignancy, unrelated (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
fall, no injury (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No